CLINICAL TRIAL: NCT00808730
Title: Role of Mitochondria in Human Bronchial Smooth Muscle Remodeling in Non Severe Asthma
Brief Title: Role of Mitochondria in Non Severe Asthma
Acronym: MITASTHME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2008/29
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Asthma
Keywords: Asthma, airway remodelling, smooth muscle, mitochondria
MeSH Terms: conditions — Asthma; Airway Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): fiberoptic fibroscopy
  Interventions: Procedure: fiberoptic fibroscopy

INTERVENTIONS:
Procedure: fiberoptic fibroscopy — Bronchial specimens will be obtained by fiberoptic bronchoscopy within 15 days after the enrolment

SUMMARY:
Asthma is a frequent disease characterized by bronchial hyperresponsiveness, inflammation and remodelling. Bronchial remodelling is an abnormal repair process that contributes to the development of poorly reversible airway narrowing. It can appear very early in the evolution of the disease and involves an increased mass of bronchial smooth muscle (BSM). The mechanism of such an increase has been related with an increase in smooth muscle cell proliferation. Recently, we have demonstrated that, BSM increased proliferation is induced by an enhanced mitochondrial biogenesis in severe asthma (T. Trian et al. J Exp Med 2007). The objective of this study is to investigate the role of smooth muscle cell mitochondria in non severe asthma

DETAILED DESCRIPTION:
Bronchial remodelling mainly involves an increased mass of bronchial smooth muscle (BSM), which is related with an increase proliferation of BSM cells. Recently, using BSM cells obtained from severe asthmatics, we have demonstrated that such an increase proliferation was induced by an activation cascade involving an abnormal calcium entry, and the subsequent activation of Calmodulin-kinase IV, PGC-1alpha, NRF-1 and mt-TFA leading to an increase mitochondrial biogenesis (T. Trian et al, J Exp Med 2007). The objective of this study is to investigate the role of BSM cell mitochondria in non severe asthma.

For this purpose, 30 non severe asthmatic adult patients (>18 yr) will be prospectively recruited from the "CHU de Bordeaux" according to the Global Initiative for Asthma (GINA) guidelines. Inclusion visit will include written informed consent, asthma control questionnaire, clinical examination, lung function testing (i.e. arterial gas, exhaled NO, plethysmography), prick tests, chest X Ray and blood sample for total IgE levels. Bronchial specimens will be obtained from all subjects by fiberoptic bronchoscopy. BSM remodelling will be evaluated by morphological analysis. Patients will be divided into 2 groups according to the presence or the absence of BSM remodelling. Using BSM cell culture, the role of mitochondria will be analyzed by electronic microscopy, confocal microscopy, immunoblotting, RT-PCR and oxygraphy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 18 years
* Diagnosis of intermittent asthma, mild persistent asthma or moderate persistent according to ATS criteria
* Forced expiratory volume in one second > 60% predicted
* Written informed consent

Exclusion Criteria:

* Smoker or former smoker (tobacco or cannabis)
* Adults protected by law
* Subjects not affiliated with social security
* Subjects during exclusion relative to another protocol or for which the annual maximum allowance of 3800 euros has been reached
* Subject with any co-morbidity (except chronic rhinitis, chronic sinusitis nasal polyps or gastro-oesophageal reflux)
* Asthma exacerbation within 6 weeks before enrolment
* Infections of the upper airway within 3 months before enrolment
* Chronic viral infections (hepatitis, HIV)
* Pregnancy or breastfeeding
* Contraindications to bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
BSM mitochondrial biogenesis assessed by the number of mitochondrial sections using electron microscopy, the porin content using western blot, and mitochondrial oxygen consumption evaluated by oxygraphy. | One bronchial fiberoptic fibroscopy within 15 days after the enrolment

SECONDARY OUTCOMES:
BSM remodelling assessed by optic microscopy and immunohistochemistry (using anti-alpha smooth muscle actin antibody). | One bronchial fiberoptic fibroscopy within 15 days after the enrolment
Transcription factors involved in mitochondrial biogenesis assessed by quantitative RT-PCR and western blot. | One bronchial fiberoptic fibroscopy within 15 days after the enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Olivier GIRODET, MCU-PH, Principal Investigator — University Hospital Bordeaux / Département de Pharmacologie, CIC - Université Victor Segalen Bordeaux 2
Locations (1):
- University Hospital Bordeaux, Hôpital Haut-Lévêque, Pessac, France

REFERENCES:
- [Background] Trian T, Benard G, Begueret H, Rossignol R, Girodet PO, Ghosh D, Ousova O, Vernejoux JM, Marthan R, Tunon-de-Lara JM, Berger P. Bronchial smooth muscle remodeling involves calcium-dependent enhanced mitochondrial biogenesis in asthma. J Exp Med. 2007 Dec 24;204(13):3173-81. doi: 10.1084/jem.20070956. Epub 2007 Dec 3. PMID 18056286
- [Derived] Girodet PO, Allard B, Thumerel M, Begueret H, Dupin I, Ousova O, Lassalle R, Maurat E, Ozier A, Trian T, Marthan R, Berger P. Bronchial Smooth Muscle Remodeling in Nonsevere Asthma. Am J Respir Crit Care Med. 2016 Mar 15;193(6):627-33. doi: 10.1164/rccm.201507-1404OC. PMID 26540234